CLINICAL TRIAL: NCT00697541
Title: A Phase II, Single-Center, Two-Way Crossover Relative Systemic Bioavailability Study of Col-118 Administered Topically as a 0.18 % Facial Gel and Brimonidine Ophthalmic Solution 0.2% Administered to the Eye in Subjects With Moderate to Severe Erythematous Rosacea
Brief Title: Systemic Bioavailability Study Of Col-118 Administered Topically as a 0.18 % Facial Gel And Brimonidine Ophthalmic Solution 0.2%
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COL-118-ROSE-202; RD.06.SPR.18126
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2014-08

CONDITIONS: Erythematous Rosacea
Keywords: erythematous rosacea; facial gel; brimonidine; ophthalmic solution
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): One 1-g application of 0.18% COL-118 facial gel (1.8 mg brimonidine) administered topically plus one drop of Advanced Eye Relief™ in each eye, once in the morning. 1 g of 0.18% COL-118 facial gel is reapplied once after four hours
  Interventions: Drug: 0.18% COL-118 facial gel (1.8 mg brimonidine); Drug: Advanced Eye Relief
- B (Active Comparator): One 1-g application of COL-118 facial gel vehicle (0.0 mg brimonidine tartrate) administered topically plus one drop of 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop) in each eye. Four hours after the first application 1-g of COL-118 facial gel vehicle (0.0 mg brimonidine) is administered topically
  Interventions: Drug: 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop); Drug: COL-118 facial gel vehicle

INTERVENTIONS:
Drug: 0.18% COL-118 facial gel (1.8 mg brimonidine) — One 1-g application of 0.18% COL-118 facial gel (1.8 mg brimonidine) administered topically plus one drop of Advanced Eye Relief™ in each eye, once in the morning. 1 g of 0.18% COL-118 facial gel is reapplied once after 4 hours
  Other Names: brimonidine
  Arms: A
Drug: 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop) — One 1-g application of COL-118 facial gel vehicle (0.0 mg brimonidine tartrate) topically plus one drop of 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop) in each eye. Four hours after the first application 1-g of COL-118 facial gel vehicle (0.0 mg brimonidine) is administered topically.
  Other Names: brimonidine tartrate/drop
  Arms: B
Drug: Advanced Eye Relief — One 1-g application of 0.18% COL-118 facial gel (1.8 mg brimonidine) administered topically plus one drop of Advanced Eye Relief™ in each eye, once in the morning. 1 g of 0.18% COL-118 facial gel is reapplied once after 4 hours
  Arms: A
Drug: COL-118 facial gel vehicle — One 1-g application of COL-118 facial gel vehicle (0.0 mg brimonidine tartrate) administered topically plus one drop of 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop) in each eye. Four hours after the first application 1-g of COL-118 facial gel vehicle (0.0 mg brimonidine) is administered topically
  Arms: B

SUMMARY:
Phase II systemic bioavailability crossover study to measure the exposure of Col-118 topical 0.18 % Facial Gel and Brimonidine Ophthalmic Solution 0.2%

DETAILED DESCRIPTION:
A double-blind, randomized, 2-way crossover, safety, pharmacokinetic/-dynamic (PK/PD) study of 0.18% COL-118 facial gel and 0.2% brimonidine ophthalmic solution administered in male and female patients with moderate to severe erythematous rosacea.

Twenty male and female subjects with moderate to severe erythematous rosacea will be randomized into 2 groups of 10 subjects.

Each group will be randomized to receive 2 treatments (Treatments A and B, in Sequence 1: A/B or Sequence 2: B/A), as follows:

Treatment A: One 1-g application of 0.18% COL-118 facial gel (1.8 mg brimonidine) administered topically plus one drop of Advanced Eye Relief™ in each eye, once in the morning. 1 g of 0.18% COL-118 facial gel is reapplied once after four hours;

Treatment B: One 1-g application of COL-118 facial gel vehicle (0.0 mg brimonidine tartrate) administered topically plus one drop of 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop) in each eye. Four hours after the first application 1-g of COL-118 facial gel vehicle (0.0 mg brimonidine) is administered topically.

There will be at least a 1-day washout between dose administrations (Period 1 and Period 2).

Blood samples for PK analysis of brimonidine levels will be collected at the following time points during Period 1 and Period 2: 0 Hour (prior to dose) and at 1, 2, 3, 4 (prior to 2nd dose), 5, 6, 7, and 8 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Clinical diagnosis of rosacea
* A score of ≥ 3 on the CEAS
* A score of ≥ 3 on the PSA
* IOP ≥ 10 mm Hg
* Non-pregnant and non-lactating females

Exclusion Criteria:

* History of hypersensitivity or allergies to any ingredient of the study drugs, unless approved by the Investigator
* Use of brimonidine prescription medications within 14 days prior to Check-in
* Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the Investigator
* Use of systemic or topical steroids applied to the face 14 days prior to Check in
* The use of any Rx or OTC products for the treatment of acne or rosacea within 14 days prior to check in
* The use of isotretinoin within 180 days prior to check in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Leyden, M.D., Principal Investigator — KGL, Inc.
Locations (1):
- KGL, Inc., Broomall, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Seq1-facial Gel+Saline Drops,Then Vehicle+Brimonidine Drops: One (1) gram of 0.18% COL-118 facial gel (1.8 mg brimonidine tartrate) administered topically plus 1 drop of Advanced Eye Relief™ (placebo ophthalmic solution) in each eye, once in the morning. One (1) gram of 0.18% COL-118 facial gel was to be reapplied once after 4 hours.
  First intervention (1 day), washout (1 day), Second intervention (1 day)
- Seq2-vehicle+Brimonidine Drops,Then Facial Gel+Saline Drops: One 1-g application of COL-118 facial gel vehicle (0.0 mg brimonidine tartrate) administered topically plus one drop of 0.2% brimonidine ophthalmic solution (0.1 mg brimonidine tartrate/drop) in each eye. Four hours after the first application 1-g of COL-118 facial gel vehicle (0.0 mg brimonidine) is administered topically
  First intervention (1 day), washout (1 day), Second intervention (1 day)
Period: Overall Study
Arm/Group | Seq1-facial Gel+Saline Drops,Then Vehicle+Brimonidine Drops | Seq2-vehicle+Brimonidine Drops,Then Facial Gel+Saline Drops
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seq1-facial Gel+Saline Drops,Then Vehicle+Brimonidine Drops | Seq2-vehicle+Brimonidine Drops,Then Facial Gel+Saline Drops | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (8.5) | 47.1 (6.7) | 45.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Systemic Concentration of Brimonidine
Description: Maximum observed plasma concentration
Time Frame: 0 Hour (prior to dose) and at 1, 2, 3, 4, 5, 6, 7, and 8 hours post-morning dose
Measure: Mean (Full Range); unit: pg/mL
Groups:
- Treatment A - COL-118 Facial Gel + Saline Drops: COL-118 facial gel + saline drops
- Treatment B - Vehicle Gel + Brimonidine Drops: Vehicle gel + brimonidine drops
Arm/Group | Treatment A - COL-118 Facial Gel + Saline Drops | Treatment B - Vehicle Gel + Brimonidine Drops
Number analyzed (Participants) | 19 | 18
pg/mL | NA (NA) [NA to NA] — After application of Brimonidine 0.18% Gel, plasma levels of brimonidine for all subjects were below the limit of quantification (< 25 pg/mL) with the exception of one single outlier value therefore no PK analysis could be performed. | NA (NA) [NA to 100] — The mean Cmax was not calculated because values were not quantifiable for 7 of 18 subjects.

2. Primary Outcome: AUC - Area Under the Curve of Brimonidine
Description: Area under the plasma concentration-time curve from 0 hour to the last measurable plasma concentration, calculated by the linear trapezoidal method
  After two topical applications of 0.18% COL-118 facial gel, plasma levels of brimonidine for all subjects were below the LoQ (25 pg/mL), with the exception of one single outlier value.
  Thus, no PK analysis could be performed for 0.18% COL-118 facial gel.
  After ocular administration of 0.2% brimonidine tartrate ophthalmic solution, quantifiable plasma concentrations of brimonidine were observed in 11 of the 18 subjects who received the brimonidine tartrate ophthalmic solution. Brimonidine rapidly appeared in plasma The mean Cmax was not calculated because values were not quantifiable for 7 of 18 subjects The mean AUC0-t also was not calculated.
Time Frame: 0 Hour (prior to dose) and at 1, 2, 3, 4, 5, 6, 7, and 8 hours post-morning dose
Measure: Mean (Full Range); unit: pg*hr/mL
Groups:
- Treatment A - COL-118 Gel + Saline Drops: COL-118 gel + saline drops
Arm/Group | Treatment A - COL-118 Gel + Saline Drops | Treatment B - Vehicle Gel + Brimonidine Drops
Number analyzed (Participants) | 19 | 18
pg*hr/mL | NA (NA) [NA to NA] — After application of Brimonidine 0.18% Gel, plasma levels of brimonidine for all subjects were below the limit of quantification (< 25 pg/mL) with the exception of one single outlier value therefore no PK analysis could be performed. | NA (NA) [NA to 471] — The mean AUC was not calculated because values were not quantifiable for 9 of 18 subjects

3. Primary Outcome: Tmax - Time to Maximum Plasma Concentration
Description: time to maximum plasma concentration
Time Frame: 0 Hour (prior to dose) and at 1, 2, 3, 4, 5, 6, 7, and 8 hours post-morning dose
Measure: Mean (Full Range); unit: Hours
Arm/Group | Treatment A - COL-118 Facial Gel + Saline Drops | Treatment B - Vehicle Gel + Brimonidine Drops
Number analyzed (Participants) | 19 | 18
Hours | NA [NA to NA] — After application of Brimonidine 0.18% Gel, plasma levels of brimonidine for all subjects were below the limit of quantification (< 25 pg/mL) with the exception of one single outlier value therefore no PK analysis could be performed. | NA [0.933 to 4.07] — After ocular administration of the 0.2% brimonidine tartrate ophthalmic solution, quantifiable plasma concentrations were observed in 11 of the 18 subjects, therefore Tmax Mean is NA.

ADVERSE EVENTS:
Groups:
- Treatment A: COL-118 gel + saline drops
- Treatment B: Vehicle gel + brimonidine drops
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 3/19 | 7/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=19) | Treatment B (N=18)
Headache (Nervous system disorders) | 3 | 5
Syncope (Nervous system disorders) | 0 | 1
pharyngolagyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days